CLINICAL TRIAL: NCT02148640
Title: A RANDOMIZED, DOUBLE-BLIND, PARALLEL-GROUP STUDY TO EVALUATE THE SAFETY AND EFFICACY OF SWITCHING FROM INNOVATOR INFLIXIMAB TO BIOSIMILAR INFLIXIMAB COMPARED WITH CONTINUED TREATMENT WITH INNOVATOR INFLIXIMAB IN PATIENTS WITH RHEUMATOID ARTHRITIS, SPONDYLOARTHRITIS, PSORIATIC ARTHRITIS, ULCERATIVE COLITIS, CROHN'S DISEASE AND CHRONIC PLAQUE PSORIASIS THE NOR-SWITCH STUDY
Brief Title: The NOR-SWITCH Study
Acronym: NOR-SWITCH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other)
Responsible Party: Principal Investigator, Tore K Kvien, Prof. Dr. Med., Diakonhjemmet Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DIA2014-01; 2014-002056-40 (EudraCT Number)
Record Dates: First submitted 2014-05-23; First posted 2014-05-28 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Rheumatoid Arthritis; Spondyloarthritis; Psoriatic Arthritis; Ulcerative Colitis; Crohn's Disease; Psoriasis Chronic
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylarthritis; Arthritis, Psoriatic; Colitis, Ulcerative; Crohn Disease | interventions — Infliximab; CT-P13

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CT-P13 (Experimental): Infusions of biosimilar infliximab (Remsima) with same dose and frequency as pre-inclusion treatment with innovator infliximab (Remicade)
  Interventions: Drug: Biosimilar infliximab
- INX (Active Comparator): Continued infusions of innovator infliximab (Remicade) with same dose and frequency as prior to inclusion
  Interventions: Drug: Innovator infliximab

INTERVENTIONS:
Drug: Innovator infliximab
  Other Names: Remicade
  Arms: INX
Drug: Biosimilar infliximab
  Other Names: Remsima
  Arms: CT-P13

SUMMARY:
The purpose of this study is to assess the safety and efficacy of switching from Remicade to the biosimilar treatment Remsima in patients with rheumatoid arthritis, spondyloarthritis, psoriatic arthritis, ulcerative colitis, Crohn's disease and chronic plaque psoriasis

ELIGIBILITY:
Inclusion Criteria:

1. A clinical diagnosis of either rheumatoid arthritis, spondyloarthritis, psoriatic arthritis, ulcerative colitis, Crohn's disease or chronic plaque psoriasis
2. Male or non-pregnant, non-nursing female
3. >18 years of age at screening
4. Stable treatment with innovator infliximab (Remicade) during the last 6 months
5. Subject capable of understanding and signing an informed consent form
6. Provision of written informed consent

Exclusion Criteria:

1. Major co-morbidities, such as severe malignancies, severe diabetic mellitus, severe infections, uncontrollable hypertension, severe cardiovascular disease (NYHA class 3 or 4) and/or severe respiratory diseases
2. Change of major co-medication during the last 2 months prior to randomization:

   RA, SpA and PsA: Initiation of systemic corticosteroids or synthetic DMARDs or other medication which according to the investigator would interfere with the stability of the disease.

   UC and CD: Initiation of systemic corticosteroids or an immunosuppressant or other medication which according to the investigator would interfere with the stability of the disease Psoriasis: Initiation of synthetic DMARDs or other medication which according to the investigator would interfere with the stability of the disease
3. Inadequate birth control, pregnancy, and/or breastfeeding
4. Psychiatric or mental disorders, alcohol abuse or other substance abuse, language barriers or other factors which makes adherence to the study protocol impossible
5. Change in treatment with innovator infliximab (Remicade) during the last 6 months due to disease related factors, not including dose/frequency adjustments due to drug concentration measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 482 (Actual)
Dates: Start 2014-10; Primary Completion 2016-06 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of disease worsening | 52 weeks
  A disease worsening in RA and PsA is defined as an increase in DAS28 of ≥ 1.2 from randomization and a minimum DAS score of 3.2.
  A disease worsening in AS/SpA is defined as an increase in ASDAS of ≥1.1 from randomization and a minimum ASDAS of 2.1.
  A disease worsening in ulcerative colitis is defined as an increase in Partial Mayo score of ≥ 3 points from randomization and a minimum partial Mayo score of ≥ 5 points.
  A disease worsening in Crohn's disease is defined as an increase in HBI of ≥ 4 points from randomization and a minimum HBI score of 7 points.
  A disease worsening in psoriasis is defined as an increase in PASI of ≥ 3 points from randomization and a minimum PASI score of 5.
  If a patient does not fulfill the formal definition, but experiences a clinically significant worsening according to both the investigator and patient and which leads to a major change in treatment this should be considered as a disease worsening but recorded separately in the CRF.

SECONDARY OUTCOMES:
Time to disease worsening | 52 weeks
Occurrence of study drug discontinuation | 52 weeks
Time to study drug discontinuation | 52 weeks
Patient's global assessment of disease activity | 52 weeks
Physicians's global assessment of disease activity | 52 weeks
Inflammation laboratory parameters | 52 weeks
  ESR and CRP for all patients, Calprotectin for UC and CD patients
Remission status according to DAS28 | 52 weeks
  For RA and PsA patients
Disease activity according to DAS28 | 52 weeks
  For RA and PsA patients
Remission status according to CDAI | 52 weeks
  For RA and PsA patients
Disease activity according to CDAI | 52 weeks
  For RA and PsA patients
Remission status according to SDAI | 52 weeks
  For RA and PsA patients
Disease activity according to SDAI | 52 weeks
  For RA and PsA patients
Remission status according to ACR/EULAR | 52 weeks
  For RA and PsA patients
Disease activity according to ACR/EULAR | 52 weeks
  For RA and PsA patients
Remission status according to ASDAS | 52 weeks
  For SpA patients
Disease activity according to ASDAS | 52 weeks
  For SpA patients
Remission status according to Partial Mayo Score | 52 weeks
  For UC patients
Disease activity according to Partial Mayo Score | 52 weeks
  For UC patients
Remission status according to Harvey-Bradshaw index | 52 weeks
  For CD patients
Disease activity according to Harvey-Bradshaw index | 52 weeks
  For CD patients
Remission status according to PASI | 52 weeks
  For psoriatic patients
Disease activity according to PASI | 52 weeks
  For psoriatic patients

OTHER OUTCOMES:
RAND SF-36 | 52 weeks
Modified Health Assessment Questionnaire (MHAQ) | 52 weeks
  Only RA, SpA and PsA patients
Inflammatory Bowel Disease Questionnaire (IBDQ) | 52 weeks
  Only UC and CD patients
Dermatology Life Quality Index (DLQI) | 52 weeks
  Only Ps patients
EQ-5D | 52 weeks
RAID | 52 weeks
  Only RA patients
PsAID | 52 weeks
  Only PsA patients
WPAI:GH | 52 weeks
  Work Productivity and Activity Impairment Questionnaire: General health
Safety and tolerability: AEs, laboratory parameters | through study completion, an average of 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tore K. Kvien, MD PhD, Principal Investigator — Diakonhjemmet Hospital
Locations (30):
- Norway (30):
  - Sørlandet Sykehus HF, Arendal
  - Ålesund Sjukehus, Helse Møre og Romsdal HF, Ålesund
  - Haukeland Universitetssjukehus Hf, Bergen
  - Haukeland Universitetssykehus, Bergen
  - Nordlandssykehuset, Bodø
  - Sykehuset Innlandet, Elverum
  - Sykehuset Østfold HF, Fredrikstad
  - Helse Førde Hf, Førde
  - Bærum Sykehus, Gjettum
  - Sykehuset Innlandet, Gjøvik
  - Sykehuset Innlandet, Hamar
  - Haugesund Sanitetsforenings Revmatismesykehus, Haugesund
  - Helse Fonna HF, Haugesund
  - Sørlandet Sykehus HF, Kristiansand
  - Helse Nord-Trøndelag, Levanger
  - Revmatismesykehuset Lillehammer, Lillehammer
  - Sykehuset Innlandet, Lillehammer
  - Akershus Universitetssykehus, Lørenskog
  - Helgelandssykehuset, Mo i Rana
  - Department of Rheumatology, Diakonhjemmet Hospital, Oslo
  - Diakonhjemmet Hospital, Oslo
  - Oslo Universitetssykehus, Rikshospitalet, Oslo
  - Oslo Universitetssykehus, Ullevål, Oslo
  - Martina Hansens Hospital, Sandvika
  - Betanien Hospital, Skien
  - Sykehuset Telemark HF, Skien
  - Universitetssykehuset i Nord-Norge, Tromsø
  - St. Olavs Hospital HF, Trondheim
  - St. Olavs Hospital, Trondheim
  - Sykehuset Vestfold, Tønsberg

REFERENCES:
- [Derived] Jorgensen KK, Goll GL, Sexton J, Bolstad N, Olsen IC, Asak O, Berset IP, Blomgren IM, Dvergsnes K, Florholmen J, Frigstad SO, Henriksen M, Hagfors J, Huppertz-Hauss G, Haavardsholm EA, Klaasen RA, Moum B, Noraberg G, Prestegard U, Rydning JH, Sagatun L, Seeberg KA, Torp R, Vold C, Warren DJ, Ystrom CM, Lundin KEA, Kvien T, Jahnsen J. Efficacy and Safety of CT-P13 in Inflammatory Bowel Disease after Switching from Originator Infliximab: Exploratory Analyses from the NOR-SWITCH Main and Extension Trials. BioDrugs. 2020 Oct;34(5):681-694. doi: 10.1007/s40259-020-00438-7. PMID 32965617
- [Derived] Goll GL, Jorgensen KK, Sexton J, Olsen IC, Bolstad N, Haavardsholm EA, Lundin KEA, Tveit KS, Lorentzen M, Berset IP, Fevang BTS, Kalstad S, Ryggen K, Warren DJ, Klaasen RA, Asak O, Baigh S, Blomgren IM, Brenna O, Bruun TJ, Dvergsnes K, Frigstad SO, Hansen IM, Hatten ISH, Huppertz-Hauss G, Henriksen M, Hoie SS, Krogh J, Midtgard IP, Mielnik P, Moum B, Noraberg G, Poyan A, Prestegard U, Rashid HU, Strand EK, Skjetne K, Seeberg KA, Torp R, Ystrom CM, Vold C, Zettel CC, Waksvik K, Gulbrandsen B, Hagfors J, Mork C, Jahnsen J, Kvien TK. Long-term efficacy and safety of biosimilar infliximab (CT-P13) after switching from originator infliximab: open-label extension of the NOR-SWITCH trial. J Intern Med. 2019 Jun;285(6):653-669. doi: 10.1111/joim.12880. Epub 2019 Apr 12. PMID 30762274
- [Derived] Jorgensen KK, Olsen IC, Goll GL, Lorentzen M, Bolstad N, Haavardsholm EA, Lundin KEA, Mork C, Jahnsen J, Kvien TK; NOR-SWITCH study group. Switching from originator infliximab to biosimilar CT-P13 compared with maintained treatment with originator infliximab (NOR-SWITCH): a 52-week, randomised, double-blind, non-inferiority trial. Lancet. 2017 Jun 10;389(10086):2304-2316. doi: 10.1016/S0140-6736(17)30068-5. Epub 2017 May 11. PMID 28502609